CLINICAL TRIAL: NCT00003284
Title: Tandem Autologous Peripheral Blood Stem Cell Transplantation (PBSCT) After High Dose Paclitaxel Followed by Ifosfamide, Carboplatin, and Etoposide (ICE) for the Treatment of Lung Cancer
Brief Title: High-Dose Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066206; CPMC-IRB-7836; CU-CAMP-017; NCI-G98-1408
Record Dates: First submitted 1999-11-01; First posted 2004-08-13 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2000-06

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; limited stage small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Filgrastim; Carboplatin; Etoposide; Ifosfamide; Paclitaxel; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose combination chemotherapy followed by peripheral stem cell transplantation in treating patients with lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate of high dose chemotherapy followed by autologous peripheral blood stem cell transplantation in the treatment of lung cancer.

OUTLINE: Patients undergo stem cell harvesting. Patients receive radiation therapy to primary site and metastatic sites, if necessary. Patients receive a high dose of paclitaxel by 24 hour continuous infusion, then stem cells are infused 72 hours later. After a 3-4 week recovery period, patients receive ifosfamide and carboplatin by daily continuous infusion on days -7, -6, -5, and -4. Etoposide is administered by continuous infusion twice daily on days -7, -6, -5, and -4. Stem cells are again infused on day 0. Filgrastim (granulocyte colony-stimulating factor; G-CSF) begins on day 0. Patients may receive radiotherapy following recovery from chemotherapy. Patients are followed weekly for the first 6 months, then periodically for at least 2 years.

PROJECTED ACCRUAL: This study will accrue 30 patients in 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically diagnosed lung cancer including the following: Relapsed limited stage small cell lung cancer (SCLC) Limited stage SCLC responding to conventional radiotherapy Extensive stage SCLC Stage IIIB and IV non-small cell lung cancer (NSCLC) Stages II-IIIA NSCLC who are unable or unwilling to undergo surgery but are acceptable candidates for high dose chemotherapy Cryopreserved peripheral blood stem cells with CD34 count greater than 2000/mm3 No untreated or uncontrolled brain metastases

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 1.5 times normal SGOT less than 1.5 times normal Renal: Creatinine clearance greater than 50 mL/min Pulmonary: Left ventricular ejection fraction greater than 45% DLCO greater than 40% Other: Not pregnant or lactating No medical or psychiatric illness preventing informed consent or intensive treatment

PRIOR CONCURRENT THERAPY: Concurrent chemotherapy allowed if no evidence of disease progression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: David G. Savage, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States